CLINICAL TRIAL: NCT01168479
Title: FLAME: Single Blind Randomized Phase III Trial to Investigate the Benefit of a Focal Lesion Ablative Microboost in Prostate Cancer
Brief Title: FLAME: Investigate the Benefit of a Focal Lesion Ablative Microboost in Prostate Cancer
Acronym: FLAME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, L.G.W. Kerkmeijer, L.G.W. Kerkmeijer, MD, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMCU-FLAME
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer; Radiotherapy; MRI
Keywords: prostate cancer; external beam radiotherapy; dose escalation; dose painting; 95Gy in 35 fractions; MRI; FLAME
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard arm (Active Comparator): The standard arm receives the current gold standard, namely 77Gy to the prostate in 35 fractions of 2.2 Gy, 5 times per week.
  Interventions: Radiation: standard arm
- FLAME boost (Experimental): In the experimental arm patients receive in addition to the current gold standard of 77 Gy to the prostate an integrated boost to the macroscopically visible tumour to reach a total dose of 95 Gy in 35 fractions of 2.7 Gy, 5 times per week.
  Interventions: Radiation: FLAME boost

INTERVENTIONS:
Radiation: FLAME boost — In the experimental arm patients receive in addition to the current gold standard of 77 Gy to the prostate an integrated boost to the macroscopically visible tumour to reach a total dose of 95 Gy in 35 fractions of 2.7 Gy, 5 times per week.
  Other Names: FLAME
  Arms: FLAME boost
Radiation: standard arm — The standard arm receives the current gold standard, namely 77Gy to the prostate in 35 fractions of 2.2 Gy, 5 times per week.
  Other Names: normal dose
  Arms: standard arm

SUMMARY:
Rationale: Dose escalation in external-beam irradiation has proven to benefit outcome in local prostate cancer. Randomized trials were performed up to doses of 78 Gy in 2 Gy fractions. Nevertheless, the five-year biochemical relapse rate still was approximately 35% in the high-dose arm. Therefore further dose escalation seems to be required. A feasibility study up to appr. 85 Gy on the entire prostate has already been performed and showed acceptable toxicity when combined with adequate position verification. Higher doses to the entire prostate are expected to increase severe toxicity. As local recurrences only occur at the site of the primary macroscopic tumour area the next step in increasing the dose should be an ablative boost to the macroscopic tumour alone, while electively irradiating the rest of the prostate to the current gold standard dose. Feasibility of this approach has been shown for an ablative dose of 95 Gy to the macroscopic tumour within the prostate.

DETAILED DESCRIPTION:
Objective:

* Primary study objective: To demonstrate the superiority of the ablative microboost dose schedule regarding 5-year biochemical no evidence of disease rate compared to the current standard of care.
* Secondary study objectives: Establish and compare the rates of treatment-related toxicity, quality of life and disease-free survival.

Study design: Single blind prospective randomized controlled phase III trial.

Study population: Patients with intermediate or high risk adenocarcinoma of the prostate. Intermediate or high risk is defined according to the Ash et al. 2000 criteria as:

* One (intermediate-risk) or more (high-risk) factors: T2, or Gleasonscore=7, or iPSA 10-20 ng/mL
* One or more (high-risk) factors: T3, or Gleasonscore >7, or iPSA >20 ng/mL

Intervention: The standard arm receives the current gold standard, namely 77Gy to the prostate in 35 fractions of 2.2 Gy, 5 times per week. In the experimental arm patients receive in addition to the current gold standard of 77 Gy to the prostate an integrated boost to the macroscopically visible tumour to reach a total dose of 95 Gy in 35 fractions of 2.7 Gy, 5 times per week.

Main study endpoint: To decrease the five-year biochemical relapse rate with at least 10%.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients will have to fill in a quality of life questionnaire before and after the radiotherapy treatments. The risk associated with the increased dose to the macroscopic tumour is an increase of toxicity and a reduction of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients scheduled for external beam radiotherapy using IMRT and fiducial marker-based position verification
* Intermediate and high risk prostate cancer, defined by Ash et al. 2000, namely:

  * One or more factors: T2, or Gleasonscore >7, or iPSA > 10 ng/mL
  * WHO score 0-2

Exclusion Criteria:

* Low risk prostate cancer, defined by Ash et al. 2000
* World Heath Organisation (WHO) score >2
* International Prostate Symptom Score (IPSS) >20
* If for any patient related reason an MRI cannot be performed
* If anticoagulation cannot be stopped temporarily regarding the implant of fiducial markers
* Previous prostatectomy (except from Trans Urethral Prostatectomy (TURP))
* TURP within 3 months from start treatment
* Previous pelvic irradiation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2009-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate the superiority of the ablative microboost dose schedule regarding 5-year biochemical no evidence of disease rate compared to the current standard of care. | Every six months for 10 years
  PSA relapse is defined by the Phoenix definition (2005) as nadir +2ng/ml.

SECONDARY OUTCOMES:
Establish and compare the rates of treatment-related toxicity. | Every six months until 10 years
  Toxicity is scored by Common Toxicity Criteria (CTC). Every grade>2 is considered severe toxicity.
quality of life | every six months until 10 year
  Quality of life is measured by: SF-36, EORTC-C30 and EORTC-PR25.
Disease specific survival | every 6 montths until 10 years
  Death with metastases is considered a death caused by the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Kerkmeijer, MD, PhD, Principal Investigator — UMC Utrecht; Uulke van der Heide, PhD, Study Director — NKI
Locations (4):
- University Hospitals Leuven, Leuven, Vlaans-Brabant, Belgium
- Netherlands (3):
  - Radboud UMC, Nijmegen, Gelderland
  - NKI-AvL, Amsterdam, North Holland
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Kowalchuk RO, Kim H, Harmsen WS, Jeans EB, Morris LK, Mullikin TC, Miller RC, Wong WW, Vargas CE, Trifiletti DM, Phillips RM, Choo CR, Davis BJ, Beriwal S, Tendulkar RD, Stish BJ, Breen WG, Waddle MR. Cost effectiveness of treatment strategies for high risk prostate cancer. Cancer. 2022 Nov 1;128(21):3815-3823. doi: 10.1002/cncr.34450. Epub 2022 Sep 7. PMID 36070558
- [Derived] Groen VH, Haustermans K, Pos FJ, Draulans C, Isebaert S, Monninkhof EM, Smeenk RJ, Kunze-Busch M, de Boer JCJ, van der Voort van Zijp J, Kerkmeijer LGW, van der Heide UA. Patterns of Failure Following External Beam Radiotherapy With or Without an Additional Focal Boost in the Randomized Controlled FLAME Trial for Localized Prostate Cancer. Eur Urol. 2022 Sep;82(3):252-257. doi: 10.1016/j.eururo.2021.12.012. Epub 2021 Dec 23. PMID 34953603
- [Derived] Kerkmeijer LGW, Groen VH, Pos FJ, Haustermans K, Monninkhof EM, Smeenk RJ, Kunze-Busch M, de Boer JCJ, van der Voort van Zijp J, van Vulpen M, Draulans C, van den Bergh L, Isebaert S, van der Heide UA. Focal Boost to the Intraprostatic Tumor in External Beam Radiotherapy for Patients With Localized Prostate Cancer: Results From the FLAME Randomized Phase III Trial. J Clin Oncol. 2021 Mar 1;39(7):787-796. doi: 10.1200/JCO.20.02873. Epub 2021 Jan 20. PMID 33471548
- [Derived] van Schie MA, Janssen TM, Eekhout D, Walraven I, Pos FJ, de Ruiter P, Kotte ANTJ, Monninkhof EM, Kerkmeijer LGW, Draulans C, de Roover R, Haustermans K, Kunze-Busch M, Smeenk RJ, van der Heide UA. Knowledge-Based Assessment of Focal Dose Escalation Treatment Plans in Prostate Cancer. Int J Radiat Oncol Biol Phys. 2020 Nov 15;108(4):1055-1062. doi: 10.1016/j.ijrobp.2020.06.072. Epub 2020 Jul 3. PMID 32629078
- [Derived] Monninkhof EM, van Loon JWL, van Vulpen M, Kerkmeijer LGW, Pos FJ, Haustermans K, van den Bergh L, Isebaert S, McColl GM, Smeenk RJ, Noteboom J, Walraven I, Peeters PHM, van der Heide UA. Standard whole prostate gland radiotherapy with and without lesion boost in prostate cancer: Toxicity in the FLAME randomized controlled trial. Radiother Oncol. 2018 Apr;127(1):74-80. doi: 10.1016/j.radonc.2017.12.022. Epub 2018 Jan 11. PMID 29336835
- [Derived] Lips IM, van der Heide UA, Haustermans K, van Lin EN, Pos F, Franken SP, Kotte AN, van Gils CH, van Vulpen M. Single blind randomized phase III trial to investigate the benefit of a focal lesion ablative microboost in prostate cancer (FLAME-trial): study protocol for a randomized controlled trial. Trials. 2011 Dec 5;12:255. doi: 10.1186/1745-6215-12-255. PMID 22141598
- See also: Click here for more information about this study: FLAME 'Multicenter Randomized Phase III Trial to Investigate the Benefit of a Focal Lesion Ablative Microboost in patients treated with External Beam Radiotherapy for Localized Prostate Cancer' — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3286435/pdf/1745-6215-12-255.pdf